CLINICAL TRIAL: NCT03078322
Title: Double-Blind, Placebo-Controlled, Phase 2 Trial to Test Efficacy and Safety of AV-101 (L-4-chlorokynurenine) as Adjunct to Current Antidepressant Therapy in Patients With Major Depressive Disorder (the ELEVATE Study)
Brief Title: AV-101 as Adjunct Antidepressant Therapy in Patients With Major Depression
Acronym: ELEVATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSG-CL 003
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AV-101 (Experimental): L-4-chlorokynurenine 1440 mg daily for 14 days
  Interventions: Drug: AV-101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-101 — Oral capsules taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Other Names: L-4-chlorokynurenine
  Arms: AV-101
Drug: Placebo — Oral capsules taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: Placebo

SUMMARY:
The study will evaluate the safety and efficacy of AV-101.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MDD, single or recurrent, and currently experiencing a MDE of at least 8 weeks in duration.
* Has a history of inadequate response to at least 1 approved antidepressant including at least 1 and no more than 3 during the current depressive episode.
* Meet the threshold on the total HAMD-17 score of > 20
* If female, a status of nonchildbearing potential or use of an acceptable form of birth control.
* Body mass index between 18 to 40 kg/m2.
* Other criteria may apply

Exclusion Criteria:

* History of bipolar disorder, schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within 6 months prior to screening.
* Women who are pregnant or breastfeeding or a positive pregnancy test at screening or baseline.
* Currently taking a prohibited adjunct therapy. Such drugs must be washed out for at least 4 weeks prior to baseline.
* Current diagnosis of moderate or severe substance use (including alcohol) disorder (abuse or dependence, as defined by DSM-5), with the exception of nicotine dependence, at screening or within 6 months prior to screening.
* In the opinion of the investigator, the subject has a significant risk for suicidal behavior
* Has received electroconvulsive therapy, or had repetitive transcranial magnetic stimulation in the current episode.
* Has received vagus nerve stimulation at any time prior to screening.
* Any current or past history of any physical condition, which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale 10-item version (MADRS-10) | 2 weeks
  Depression questionnaire

SECONDARY OUTCOMES:
Time course of improvement including response rates | 2 weeks
  50% improvement on MADRS-10
Safety and tolerability will be assessed by incidence of adverse events (AEs) | 2 weeks
  Also include EKG, labs etc.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - VistaGen Investigational Site, Garden Grove, California
  - VistaGen Investigational Site, Los Angeles, California
  - VistaGen Investigational Site, National City, California
  - VistaGen Investigational Site, Oakland, California
  - VistaGen Investigational Site, San Diego, California
  - VistaGen Investigational Site, Temecula, California
  - VistaGen Investigational Site, Fort Myers, Florida
  - VistaGen Investigational Site, Jacksonville, Florida
  - VistaGen Investigational Site, Atlanta, Georgia
  - VistaGen Investigational Site, Augusta, Georgia
  - VistaGen Investigational Site, Hoffman Estates, Illinois
  - VistaGen Investigational Site, Lake Charles, Louisiana
  - VistaGen Investigational Site, Gaithersburg, Maryland
  - VistaGen Investigational Site, St Louis, Missouri
  - VistaGen Investigational Site, New York, New York
  - VistaGen Investigational Site, Rochester, New York
  - VistaGen Investigational Site, Dayton, Ohio
  - VistaGen Investigational Site, Oklahoma City, Oklahoma
  - VistaGen Investigational Site, Media, Pennsylvania
  - VistaGen Investigational Site, Houston, Texas
  - VistaGen Investigational Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No